CLINICAL TRIAL: NCT00285571
Title: Dietary Variety vs Dietary Fat Effects on Energy Intake
Brief Title: Dietary Variety Versus Dietary Fat Effects in Energy Intake
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DK62400 (completed 2007)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Healthy

INTERVENTIONS:
Behavioral: Controlled Feeding Intervention

SUMMARY:
The relative importance of dietary patterns vs. macronutrient composition in affecting energy intake and body weight remains uncertain. In this study we propose to investigate the relative effects of dietary variety vs dietary fat on voluntary energy intake in adults. We will quantify and compare the effects of typical ranges of variety & fat intakes in the American diet on voluntary energy intake. The primary hypotheses to be tested are 1)an increasing availability of entree/side/snack/dessert variety offered will significantly increase voluntary energy intake in a dose-response fashion when other dietary factors known to influence energy intake are held constant. 2)The separate effects of dietary variety & dietary fat on energy intake will be similar.

We anticipate that the results of this investigation will lead to a greater understanding of the relative importance of eating patterns versus macronutrient composition in the etiology of obesity, and more specifically, dietary variety versus dietary fat in determining energy intake. More importantly, it will help lay a foundation for improved dietary recommendations concerning weight loss and prevention of excess weight gain in adulthood.

DETAILED DESCRIPTION:
The relative importance of dietary patterns vs. macronutrient composition in affecting energy intake and body weight remains uncertain. In this study we propose to investigate the relative effects of dietary variety vs dietary fat on voluntary energy intake in adults. We will quantify and compare the effects of typical ranges of variety & fat intakes in the American diet on voluntary energy intake. The primary hypotheses to be tested are 1)an increasing availability of entree/side/snack/dessert variety offered will significantly increase voluntary energy intake in a dose-response fashion when other dietary factors known to influence energy intake are held constant. 2)The separate effects of dietary variety & dietary fat on energy intake will be similar.

We anticipate that the results of this investigation will lead to a greater understanding of the relative importance of eating patterns versus macronutrient composition in the etiology of obesity, and more specifically, dietary variety versus dietary fat in determining energy intake. More importantly, it will help lay a foundation for improved dietary recommendations concerning weight loss and prevention of excess weight gain in adulthood

ELIGIBILITY:
Inclusion Criteria: Healthy adults age 18-5 y with BMI 20-35 kg/m

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in energy intake at two weeks.

SECONDARY OUTCOMES:
Two week changes in body weight, fat, taste preferences, nutrient composition of self-selected dietary intake, eating patterns of self-selected dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Megan McCrory, PhD, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University, Kenmore, Washington, United States